CLINICAL TRIAL: NCT00500136
Title: The Effects of Religion and Motivation on Medical Decision Making: A Terror Management Approach
Brief Title: The Psychosocial Effect of Thoughts of Personal Mortality on Cardiac Risk Assessment by Medical Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jamie Arndt, Principal Investigator, University of Missouri-Columbia
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: 1078398; R01CA096581 (NIH)
Record Dates: First submitted 2007-07-10; First posted 2007-07-12 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-10

CONDITIONS: Prejudice
Keywords: bias
MeSH Terms: conditions — Prejudice

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: mortality salience

SUMMARY:
This study was designed to examine if provoking thoughts of mortality among medical students can influence cardiac risk assessments depending on the religion of the target patient.

DETAILED DESCRIPTION:
This study was designed to examine whether and how provoking thoughts of mortality among medical students can influence cardiac risk assessments depending on the religion of the target patient.

ELIGIBILITY:
Inclusion Criteria:

* medical students

Exclusion Criteria:

* non-medical students

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2007-01; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Responses on a scale of 0-100 to each of three cardiac risk questions | immediate

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Arndt, PhD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Greenberg J, Solomon S, Pyszczynski T. Terror management theory of self-esteem and cultural worldviews: Empirical assessments and conceptual refinements. In: Zanna MP, ed. Advances in Experimental Social Psychology. San Diego, CA: Academic Press; 1997:61-139.